CLINICAL TRIAL: NCT06303544
Title: More Outside Your Door (MOYD): a Multilevel Intervention Promoting Traditional Diet and Physical Activity to Decrease Risk of Obesity in Alaska Native (AN) Preschoolers
Brief Title: More Outside Your Door: a Diet/physical Activity Intervention to Decrease Risk of Obesity in Alaska Native Preschoolers
Acronym: MOYD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alaska Native Tribal Health Consortium (Other)
Collaborators: Washington State University (Other); University of Alaska Anchorage (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: R01HL168853 (NIH)
Record Dates: First submitted 2023-11-07; First posted 2024-03-12 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Child Obesity
Keywords: Head Start, CBPR
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Wedge design using repeated cross sectional samples of Head Start preschool students
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Wedge 1 (Experimental): Four villages of 12 will be randomized into Wedge 1. Four of the remaining 8 villages will be randomized to Wedge 2. The remaining 4 villages will be Wedge 3.
  Interventions: Behavioral: Wedge 1
- Wedge 2 (No Intervention): While Wedge 1 is undergoing intervention, Wedges 2 & 3 will act as controls.
- Wedge 3 (No Intervention): While Wedge 1 is undergoing intervention, Wedges 2 & 3 will act as controls.

INTERVENTIONS:
Behavioral: Wedge 1 — Wedge1 will receive intervention consisting of culturally based physical activity module, built environment, community healthy lifestyle promotion
  Arms: Wedge 1

SUMMARY:
The preschool age is a crucial period of growth and an optimal time to begin to establish healthy eating and physical activity habits leading to better food and activity choices into adulthood, thereby minimizing risk for obesity-related diseases and decreasing the cardiometabolic disparities in this Indigenous population. More Outside Your Door is a multi-level, randomized, stepped-wedge intervention trial designed to reduce the disparity of childhood obesity in Yup'ik Alaska Native children by increasing the proportion of nutrient-dense traditional and traditional-like foods offered and increasing physical activity, particularly outdoor activities related to traditional Yup'ik subsistence and lifestyle practices. This 5-year intervention trial targeting 3-5 year olds is conducted in partnership with Rural Action Community Action Program Head Start programs in 12 rural Alaskan communities, where each site is assigned annually to a wedge group to receive either a community-altered culturally-tailored 8-month traditional foods and activities curriculum intervention or the standard regional Head Start program intervention.

DETAILED DESCRIPTION:
The Rural Alaska Community Action Program (RurAL CAP), which administers Head Start schools in rural Alaska, reports that 68% of Alaska Native children ages 3 to 5 years are overweight and 43% are obese. Diet, physical activity, and sleep hygiene are primary risk factors for childhood obesity, a risk factor for cardiometabolic diseases later in life. Notably, subclinical cardiovascular pathology can be detected as early as 3 years of age. Once living off the land and sea, Alaska Native (AN) people have suffered decades of colonization and in-migration, which have interfered with traditional food consumption, signaling a striking change in local food systems. Diet and physical activity are prime targets for early intervention, as taste preferences and exercise habits established in childhood forge lifelong adherence. Thus, investigators have designed More Outside Your Door, a multilevel intervention, which at the individual level builds on prior efforts to promote traditional diet and activities to decrease risk for obesity in Alaska Native preschoolers. At the family level, MOYD provides feedback to parents about their child's health screenings; at the school level, it features traditional foods, outdoor traditional physical activities, and a culturally centered curriculum. At the community level, it offers resources to improve the built environment for safe outdoor play that invites all community members to participate. In partnership, the Alaska Native Tribal Health Consortium, RurAL CAP, and collaborators will refine and test the effectiveness of MOYD at 12 Head Start preschools in the Yukon-Kuskokwim region: (1) investigators will use qualitative methods with Head Start staff, parents, and community Elders to optimally tailor MOYD for southwest Alaska communities; (2) investigators will conduct a stepped-wedge group-randomized trial to test its effect on children's diet, physical activity (PA), body mass index (BMI), and other risk factors for obesity-related chronic disease over three years. Primary outcomes are diet (classroom meals, actigraphy-based physical activity, and body mass index. Secondary outcomes include individual child level measures of hemoglobin levels and educational and developmental progress; parent report of diet, activity, and sleep at home; and measures of traditional foods/sugar-sweetened/processed foods by carbon and nitrogen stable isotope ratios using fingernail clippings. Investigators will also measure outcomes at the school level (classroom meals, outdoor time) and community level (objective data on use of play space). (3) Investigators will conduct a process evaluation using the RE-AIM framework. The Specific Aims are to (1) conduct preschool staff and parent/elder workgroups to refine the MOYD intervention for optimal effectiveness for obesity prevention among AN preschool children; (2) test the effectiveness of MOYD on a) diet, PA, outdoor time, and BMI; and b) improving other clinical and behavioral risk factors for obesity-related chronic disease in preschool children; and (3) Implement the RE-AIM framework to evaluate dissemination and implementation of the MOYD intervention in Head Start programs.

ELIGIBILITY:
Inclusion Criteria:

* parent who identifies as Alaska Native (AN)
* parental consent
* enrolled in preschool in one of the12 participating Head Start programs
* present at school for health screenings

Exclusion Criteria:

* lack of parental consent
* does not have a parent who is AN

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
BMI | 3 years
  Body mass index (kg/m2)
Physical activity | 3 years
  Measured via accelerometers (minutes)
Outdoor time | 3 years
  Time (minutes) spent outdoors by children
Sleep quality | 3 years
  Hours of sleep measured by survey
Fingernail nitrogen & carbon stable isotope ratios | 3 years
  Measurements of traditional food intake and added sugar intake

CONTACTS AND LOCATIONS:
Locations (1):
- Alaska Native Tribal Health Consortium, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No
Any shared data will be deidentified.